CLINICAL TRIAL: NCT04466618
Title: To Determine the Effect of Endogenous GLP-1 Secretion on Islet Function in People With and Without Type 2 Diabetes
Brief Title: Endogenous GLP-1 Secretion on Islet Function in People With and Without Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Adrian Vella (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Adrian Vella, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20-003993; R01DK126206 (NIH)
Record Dates: First submitted 2020-06-30; First posted 2020-07-10 (Actual); Results first posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Healthy; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sodium Chloride; soybean oil, phospholipid emulsion; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Saline (Placebo Comparator): Saline infusion
  Interventions: Biological: Saline
- Exendin-9,39 (Active Comparator): Exendin-9,39 infusion
  Interventions: Biological: Exendin-9,39
- Saline + Intralipid/Heparin (Active Comparator): Induction of acute insulin resistance during Saline infusion
  Interventions: Biological: Saline + Intralipid/Heparin
- Exendin-9,39 + Intralipid/Heparin (Active Comparator): Induction of acute insulin resistance during Exendin-9,39 infusion
  Interventions: Biological: Exendin-9,39 + Intralipid/Heparin

INTERVENTIONS:
Biological: Saline — Saline infused during the study
  Arms: Saline
Biological: Exendin-9,39 — Exendin-9,39 infused during the study
  Arms: Exendin-9,39
Biological: Saline + Intralipid/Heparin — Saline infused during acute insulin resistance
  Arms: Saline + Intralipid/Heparin
Biological: Exendin-9,39 + Intralipid/Heparin — Exendin-9,39 infused during acute insulin resistance
  Arms: Exendin-9,39 + Intralipid/Heparin

SUMMARY:
GLP-1 is a hormone made by the body that promotes the production of insulin in response to GLP-1 is produced within the islets expressing prohormone convertase 1/3eating. However, there is increasing evidence that this hormone might help support the body's ability to produce insulin when diabetes develops. The purpose of this study is to determine the effect of endogenous GLP-1 secretion on insulin secretion in people with and without type 2 diabetes.

DETAILED DESCRIPTION:
Accumulating evidence suggests that in rodents and humans GLP-1 is synthesized within islets and may act locally in a paracrine fashion. Indeed, mice with genetic loss of intra-islet GLP-1 exhibit decreased insulin secretion and impaired response to metabolic stressors. 'Pancreatic' GLP-1 may contribute to the effects of DPP-4 inhibitors in rodents and humans. Antagonism of GLP1R with exendin-9,39 during fasting impairs the islet cell response to an I.V. glucose challenge. Islet GLP-1 content is increased in T2DM and in islets from non-diabetic humans exposed to hyperglycemia and Free Fatty Acids. These observations imply that paracrine GLP-1 secretion supports islet function in the presence of glucolipotoxicity. In this experiment we will examine the role of endogenous GLP-1 secretion in people with and without T2DM and during β-cell stress induced by FFA elevation.

ELIGIBILITY:
Inclusion criteria - non-diabetic subjects:

* Weight-stable, non-diabetic subjects

Exclusion Criteria - non-diabetic subjects:

* Age < 25 or > 65 years (to avoid studying subjects who could have latent type 1 diabetes, or the effects of age extremes in subjects with normal or impaired fasting glucose).
* HbA1c ≥ 6.5%
* Use of glucose-lowering agents.
* For female subjects: positive pregnancy test at the time of enrollment or study
* History of prior upper abdominal surgery such as adjustable gastric banding, pyloroplasty and vagotomy.
* Active systemic illness or malignancy.
* Symptomatic macrovascular or microvascular disease.

Inclusion criteria - diabetic subjects:

* Weight-stable, diabetic subjects treated with diet and lifestyle alone or with metformin monotherapy

Exclusion Criteria - diabetic subjects:

* Age < 25 or > 65 years (to avoid studying subjects who could have latent type 1 diabetes, or the effects of age extremes in subjects with normal or impaired fasting glucose).
* Use of any glucose-lowering agent other than metformin.
* 2 or more fasting glucose values > 250mg/dl on medication or after medication withdrawal.
* Unwillingness or inability to withdraw medication for three weeks prior to, and for the duration of the study.
* For female subjects: positive pregnancy test at the time of enrollment or study
* History of prior upper abdominal surgery such as adjustable gastric banding, pyloroplasty and vagotomy.
* Active systemic illness or malignancy.
* Symptomatic macrovascular or microvascular disease.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Welch AA, Farahani RA, Egan AM, Laurenti MC, Zeini M, Vella M, Bailey KR, Cobelli C, Dalla Man C, Matveyenko A, Vella A. Glucagon-like peptide-1 receptor blockade impairs islet secretion and glucose metabolism in humans. J Clin Invest. 2023 Nov 15;133(22):e173495. doi: 10.1172/JCI173495. PMID 37751301
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-diabetic Subjects: Saline: Saline infused during the study
  Exendin-9,39: Exendin-9,39 infused during the study
  In a subset an additional 2 arms: -
  Saline + Intralipid/Heparin: Saline infused during acute insulin resistance
  Exendin-9,39 + Intralipid/Heparin: Exendin-9,39 infused during acute insulin resistance
- Subjects With Type 2 Diabetes: Saline: Saline infused during the study
  Exendin-9,39: Exendin-9,39 infused during the study
Period: Overall Study
Arm/Group | Non-diabetic Subjects | Subjects With Type 2 Diabetes
Started | 12 | 11
Completed | 12 | 10
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- No Diabetes: Subjects without Diabetes
- Type 2 Diabetes: Subjects with Type 2 Diabetes
- Total: Total of all reporting groups
Arm/Group | No Diabetes | Type 2 Diabetes | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (8) | 58 (5) | 56 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 4 | 3 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Fasting Glucagon in the Presence or Absence of Exendin-9,39
Description: Concentrations of glucagon Measured by immunoassay over the -30 to 0 minutes of study.
  On one study day subjects received saline, on the other exendin-9,39. The infusion commenced at -120 minutes.
Time Frame: Average concentration over the -30 to 0 minutes of study
Population: 1 patient with type 2 diabetes did not complete one study secondary to loss of IV access
Measure: Mean (Standard Error); unit: pmol/l
Arm/Group | No Diabetes | Type 2 Diabetes
Number analyzed (Participants) | 12 | 11
pmol/l
  Saline: number analyzed (Participants) | 12 | 10
  Saline | 7.4 (1.2) | 7.9 (0.3)
  Exendin 9-39 | 7.8 (1.1) | 10.2 (0.3)

ADVERSE EVENTS:
Time Frame: The 3 months of participation
Groups:
- Non-diabetic Subjects Saline: Subjects without Diabetes and Saline infused.
- Non-diabetic Subjects Exendin-9,39: Subjects without Diabetes and Exendin-9,39 infused.
- Non-diabetic Subjects Saline + Intralipid/Heparin: Subjects without Diabetes and Saline + Intralipid/Heparin infused.
- Non-diabetic Subjects Exendin-9,39 + Intralipid/Heparin:: Subjects without Diabetes and Exendin-9,39 + Intralipid/Heparin infused.
- Type 2 Diabetes Saline: Subjects with Type 2 Diabetes and Saline infused.
- Type 2 Diabetes Exendin-9,39: Subjects with Type 2 Diabetes and Exendin-9,39 infused.
Arm/Group | Non-diabetic Subjects Saline | Non-diabetic Subjects Exendin-9,39 | Non-diabetic Subjects Saline + Intralipid/Heparin | Non-diabetic Subjects Exendin-9,39 + Intralipid/Heparin: | Type 2 Diabetes Saline | Type 2 Diabetes Exendin-9,39
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 1/11 | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-diabetic Subjects Saline (N=12) | Non-diabetic Subjects Exendin-9,39 (N=12) | Non-diabetic Subjects Saline + Intralipid/Heparin (N=12) | Non-diabetic Subjects Exendin-9,39 + Intralipid/Heparin: (N=12) | Type 2 Diabetes Saline (N=11) | Type 2 Diabetes Exendin-9,39 (N=11)
Hyperglycemia (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — one patient presented with hyperglycemia on the morning of the study
IV access loss (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT04466618/Prot_SAP_000.pdf